CLINICAL TRIAL: NCT02416102
Title: Effect of Losartan on Airway Mucociliary Dysfunction in Patients With COPD and Chronic Bronchitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Flight Attendant Medical Research Institute (Other)
Responsible Party: Principal Investigator, Rafael Calderon Candelario, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20140722; R01HL133240 (NIH); R01HL139365 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-04-14 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: COPD; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy non-smokers (Active Comparator): 10 healthy non-smokers will receive 50 mg of Losartan for 4 consecutive weeks followed by 100 mg of Losartan for 4 consecutive weeks.
  Interventions: Drug: Losartan 50 mg; Drug: Losartan 100 mg
- Smokers without COPD (Experimental): 10 smokers without COPD will receive 50 mg of Losartan for 4 consecutive weeks followed by 100 mg of Losartan for 4 consecutive weeks.
  Interventions: Drug: Losartan 50 mg; Drug: Losartan 100 mg
- Ex-smokers with COPD (Experimental): 10 ex-smokers with COPD will receive 50 mg of Losartan for 4 consecutive weeks followed by 100 mg of Losartan for 4 consecutive weeks.
  Interventions: Drug: Losartan 50 mg; Drug: Losartan 100 mg

INTERVENTIONS:
Drug: Losartan 50 mg — 50 mg Losartan taken orally once daily for 4 consecutive weeks.
  Other Names: Cozaar
Drug: Losartan 100 mg — 50 mg Losartan taken orally twice daily for 4 consecutive weeks.
  Other Names: Cozaar

SUMMARY:
The purpose of this study is to evaluate the effect of Losartan on cigarette smoke-induced lung injury in smokers and ex-smokers with and without chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill one of the group definitions above
2. Age between 35 and 75 years old
3. Clinical diagnosis of chronic bronchitis, defined as productive cough for at least 3 months per year for at least two consecutive years
4. Stable maintenance of all current medication therapy for 3 months, including ARBs for treated groups

Exclusion criteria

1. Current therapy with Angiotensin-converting-enzyme (ACE) inhibitor,or Intolerance to Angiotensin II receptor blockers (ARB)
2. Women of child bearing potential
3. Current use of nonsteroidal antiinflammatory drugs or potassium supplementation, treatment with aliskiren, anticoagulation
4. COPD exacerbation requiring treatment within 6 weeks of the screening visit
5. Oral corticosteroid use within 6 weeks of the screening visit
6. Significant hypoxemia (oxygen saturation <90% on room air), chronic respiratory failure by history (pCO2 > 45 mmHg) and forced expiratory volume in 1 second (FEV1) below 40%, clinical evidence of cor pulmonale
7. Untreated arterial hypertension (systolic blood pressure >140 mm Hg, diastolic blood pressure > 90 mm Hg)
8. Ability to understand and willingness to sign consent documents
9. Blood pressure less than 100 mm Hg systolic or 70 mm Hg diastolic while standing at the screening visit
10. Cardiac, renal, hepatic (LFTs > 3x normal upper limit), neurological, psychiatric, endocrine or neoplastic diseases that are at the discretion of the investigator, to interfere with participation in study
11. History of renal artery stenosis
12. Concomitant airway disorders other than COPD and chronic bronchitis, such as bronchiectasis and asthma (history and reversible airflow obstruction by American Thoracic Society (ATS) criteria)
13. History of pulmonary malignancies, and any other malignancies in the last 5 years
14. History of thoracic surgery.
15. Acute pulmonary exacerbation within 6 weeks from the Screening Visit.
16. Subjects with no airflow obstruction by spirometry but with a decrease in diffusing capacity of lung for carbon monoxide(DLco) possibly indicating emphysema.
17. Significant exposure to environmental tobacco smoke or atmospheric or occupational pollutants
18. Urine pregnancy positive test at the Screening Visit.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Calderon, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Non-smokers: 10 healthy non-smokers will receive 50 mg of losartan for 4 weeks followed by 100 mg of losartan for 4 weeks
  Losartan 50 mg: 50 mg once daily (QD) for 4 weeks
  losartan 100 mg: 50 mg twice daily (BID) for 4 weeks
- Smokers Without COPD: 10 smokers without Chronic Obstructive Pulmonary Disease (COPD) will receive 50 mg of losartan for 4 weeks followed by 100 mg of losartan for 4 weeks
  Losartan 50 mg: 50 mg QD for 4 weeks
  losartan 100 mg: 50 mg BID for 4 weeks
- Ex-smokers With COPD: 10 ex-smokers with COPD will receive 50 mg of losartan for 4 weeks followed by 100 mg of losartan for 4 weeks
  Losartan 50 mg: 50 mg QD for 4 weeks
  losartan 100 mg: 50 mg BID for 4 weeks
Period: Overall Study
Arm/Group | Healthy Non-smokers | Smokers Without COPD | Ex-smokers With COPD
Started | 16 | 15 | 0
Completed | 7 | 7 | 0
Not Completed | 9 | 8 | 0

BASELINE CHARACTERISTICS:
Population: There was a difficulty in recruitment ex-smokers with COPD prior to study termination
Groups:
- Healthy Non-smokers: 10 healthy non-smokers will receive 50 mg of losartan for 4 weeks followed by 100 mg of losartan for 4 weeks
  Losartan 50 mg: 50 mg QD for 4 weeks
  losartan 100 mg: 50 mg BID for 4 weeks
- Smokers Without COPD: 10 smokers without COPD will receive 50 mg of losartan for 4 weeks followed by 100 mg of losartan for 4 weeks
  Losartan 50 mg: 50 mg QD for 4 weeks
  losartan 100 mg: 50 mg BID for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Healthy Non-smokers | Smokers Without COPD | Ex-smokers With COPD | Total
Number analyzed (Participants) | 16 | 15 | 0 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 0 | 30
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 0 | 21
  Male | 3 | 7 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 0 | 26
  Not Hispanic or Latino | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 13 | 9 | 0 | 22
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 3 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Nasal Potential Difference (NPD).
Description: NPD were assessed from nasal cells collected using sterile cytology brushes.
Time Frame: Baseline, 8 weeks
Population: Nasal sample data for all participants were not available as the readings were uninterpretable and not further analyzed.
Arm/Group | Healthy Non-smokers | Smokers Without COPD | Ex-smokers With COPD
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in IL-8 Concentrations
Description: Interleukin (IL)-8 concentrations were analyzed from samples on nasal lavage
Time Frame: Baseline, 8 weeks
Population: No participants were recruited in the Ex-Smokers with COPD due to difficulty in recruitment prior to study termination. Only 5 participants were analyzed for the Healthy Non-Smokers and Smokers without COPD arms as only 5 in each group had complete sets of samples that could be analyzed due to bad quality/quantity available.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Non-smokers | Smokers Without COPD | Ex-smokers With COPD
Number analyzed (Participants) | 5 | 5 | 0
pg/mL | 2867 (1685) | 4676 (1948) |

3. Secondary Outcome: Percent Change in TGF-ß mRNA Expression
Description: Transforming Growth Factor (TGF)-ß messenger ribonucleic acid (mRNA) expression were analyzed from nasal cells samples.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change in mRNA expression
Arm/Group | Healthy Non-smokers | Smokers Without COPD | Ex-smokers With COPD
Number analyzed (Participants) | 5 | 5 | 0
percentage change in mRNA expression | -51 (31) | -23 (70) |

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Only treatment-emergent Adverse Events will be reported as per treating physician discretion.
Arm/Group | Healthy Non-smokers | Smokers Without COPD | Ex-smokers With COPD
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/0
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02416102/Prot_SAP_000.pdf